CLINICAL TRIAL: NCT05282654
Title: Real-time Symptom Monitoring Using ePROs to Prevent Adverse Events During Care Transitions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: RAND (Other)
Responsible Party: Principal Investigator, Anuj K. Dalal, MD, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021P002593
Record Dates: First submitted 2022-02-11; First posted 2022-03-16 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Multiple Chronic Conditions; Adverse Event
Keywords: Digital Health; Patient Reported Outcomes; Symptom Monitoring; Predictive Model; Care Transitions; Post Acute Care
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: Baseline, pre-implementation period (usual care arm 1) and main trial (RCT) period (usual care arm 2 and intervention/experimental arm 3)
Who Masked: Investigator, Outcomes Assessor
Masking Description: During main trial (post-implementation period), study investigators, outcomes assessor will be masked to randomization status of all participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Arm 1) (No Intervention): During the 18-month Baseline Period (Arm 1, n=450) patients will be enrolled and receive usual care to develop the initial predictive model.
- Usual Care (Arm 2) (No Intervention): During the 30-month Main Trial (RCT) Period, patients will be randomized to usual care (Arm 2, n=425). Data collection for post-discharge AE determination will occur during both periods.
- Intervention (Arm 3) (Experimental): During the 30-month Main Trial (RCT) Period, patients will be randomized to the intervention (Arm 3, n=425). Data collection for post-discharge AE determination will occur during both periods.
  Interventions: Behavioral: ePRO Application

INTERVENTIONS:
Behavioral: ePRO Application — The intervention consists of a patient portal, EHR-integrated web-app to communicate risk of post-discharge adverse events using patient-reported outcome questionnaires, discharge preparation checklist during hospitalization. After discharge, the intervention will provide real-time symptom monitoring using ePROs and facilitate communication with clinicians based on prediction model-informed ePRO score trends exceeding escalation thresholds.
  Arms: Intervention (Arm 3)

SUMMARY:
This study aims to predict and minimize post-discharge adverse events (AEs) during care transitions through early identification and escalation of patient-reported symptoms to inpatient and ambulatory clinicians by way of predictive algorithms and clinically integrated digital health apps. We will (1) develop and prospectively validate a predictive model of post-discharge AEs for patients with multiple chronic conditions (MCC); (2) combine, adapt, extend, and iteratively refine our EHR-integrated digital health infrastructure in a series of design sessions with patient and clinician participants; (3) conduct a RCT to evaluate the impact of ePRO monitoring on post-discharge AEs for MCC patients discharged from the general medicine service across Brigham Health; and (4) use mixed methods to evaluate barriers and facilitators of implementation and use as we develop a plan for sustainability, scale, and dissemination.

DETAILED DESCRIPTION:
Adverse events (AE) during care transitions range from 19-28% and may lead to readmissions, representing an ongoing threat to patient safety. Early identification and escalation of patient-reported symptoms to inpatient and ambulatory clinicians is critical, especially for patients with multiple chronic conditions (MCC). Clinically integrated digital health apps have the potential to more accurately predict post-discharge AEs and improve communication for patients, their caregivers, and the care team. Such tools can provide individualized risk assessments of AEs by systematically collecting relevant patient-reported outcomes (PROs) and leveraging standardized application programming interfaces (API) to combine them with electronic health record (EHR) data. While patient-reported outcomes (PROs) are increasingly used in ambulatory settings, their use for real-time symptom monitoring and escalation during transitions from the hospital is novel and potentially transformative-by both empowering patients to better understand their individualized risks of post-discharge AEs, and improving monitoring while transitioning out of the hospital. Our proposed intervention is grounded in evidence-based frameworks for care transitions, and scaling and spread of digital health tools. To inform our intervention, we propose developing and validating a predictive model of post-discharge AEs for 450 MCC patients using relevant PRO questionnaires and electronic health record (EHR) derived variables during our baseline pre-implementation period. Simultaneously, we will combine, adapt, extend, and refine our previously developed EHR-integrated hospital and ambulatory-focused digital health infrastructure to support MCC patients in real-time symptom monitoring using PROs when transitioning out of the hospital. Our intervention uses interoperable, data exchange standards and APIs to seamlessly integrate with existing vendor patient portal offerings, thereby addressing critical gaps and supporting the complete continuum of care. Our multidisciplinary team uses principles of user-centered design and agile software development to rapidly identify, design, develop, refine, and implement requirements from patients and clinicians. Our team will rigorously evaluate this intervention in a large-scale randomized controlled trial of 850 in which we compare our real-time symptom monitoring intervention (425) to usual care (425) for patients with MCCs transitioning out of the hospital. Finally, we will conduct a robust mixed methods evaluation to generate new knowledge and best practices for disseminating, implementing, and using this interoperable intervention at similar institutions with different EHR vendors

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* Hospitalized on the general medicine services at Brigham and Women's Hospital or Brigham and Women's Faulkner Hospital for at least 24 hours
* Have a discharge status of home, home with services, or facility
* English-speaking patients or their English-speaking legally designated healthcare proxy or next of kin (i.e., a family caregiver)
* Non-English-speaking patients who have an English-speaking legally designated healthcare proxy or next of kin (i.e., a family caregiver)
* Two or more chronic conditions: Anxiety, Asthma*, Arthritis (Osteoarthritis, Rheumatoid), Atrial Fibrillation, Cancer*, Cerebral vascular accident, Chronic kidney disease*, Chronic obstructive pulmonary disease (COPD)*, Cirrhosis, Coronary artery disease/Ischemic heart disease, Dementia, Depression, Diabetes mellitus*, End-stage renal disease*, Heart failure*, Hepatitis B, C*, HIV/AIDs, Hyperlipidemia, Hypertension, Inflammatory bowel disease, Osteoporosis, Sickle cell disease, Substance abuse (Alcohol/Opioid)

Exclusion Criteria:

* Less than 18 years of age
* Less than two chronic conditions
* Hospitalized less than 24 hours
* No identifiable healthcare proxy or next of kin (i.e., a family caregiver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Actual adverse events (AEs) | Up to 30-days after discharge from index hospitalization
  The number of actual AEs during the 30-day post-discharge period
Actual preventable adverse events (AEs) | Up to 30-days after discharge from index hospitalization
  The number of actual AEs during the 30-day post-discharge period

SECONDARY OUTCOMES:
Potential adverse events (AEs) | Up to 30-days after discharge from index hospitalization
  The number of new or worsening symptoms reported by the patient
Post-discharge healthcare utilization events (hospital readmissions) | Up to 30-days after discharge from index hospitalization
  Hospital readmissions
Post-discharge healthcare utilization (ambulatory events) | Up to 30-days after discharge from index hospitalization
  Composite of unanticipated ambulatory, urgent care, ED visits

OTHER OUTCOMES:
Time to actual AE | Up to 30-days after discharge from index hospitalization
  The number of days until first AE detected
Time to potential AE | Up to 30-days after discharge from index hospitalization
  The number of days until first potential AE detected

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Dalal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts